CLINICAL TRIAL: NCT04122378
Title: A Pilot Study of Acupuncture for the Treatment of Pain in Sickle Cell Disease
Brief Title: Acupuncture for Pain in Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deepika Darbari (Other)
Responsible Party: Sponsor-Investigator, Deepika Darbari, Associate Professor of Pediatrics, Division of Hematology, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00010719
Record Dates: First submitted 2019-10-02; First posted 2019-10-10 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2022-07

CONDITIONS: Sickle Cell Disease
Keywords: Pain, Acupuncture
MeSH Terms: conditions — Anemia, Sickle Cell; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Proposed study is a feasibility study of acupuncture therapy in patients with SCD admitted for management of acute pain. The primary goal of proposed study is to determine (1) if acupuncture is acceptable modality for management of pain in patients with SCD. The investigators will also explore (2) if acupuncture improves pain outcomes in SCD and (3) if use of acupuncture is associated with modulation of cytokines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Acupuncture will be provided up to once daily for one or more days till the day of discharge or 5 days, whichever occurs first. Patients will continue to receive their standard pain management regime including IV opioids, ketorolac and fluids. Minimum number of sessions received by the acupuncture group will be one.
  Interventions: Other: acupuncture
- Control Arm (No Intervention): Standard of care for SCD patients who are hospitalized for acute pain and typically includes IV opioids, ketorolac and fluids.

INTERVENTIONS:
Other: acupuncture — The acupuncture will be provided by the licensed acupuncturist using standard methods.
  Arms: Treatment Arm

SUMMARY:
Sickle cell disease (SCD) is the most common genetic disorder in the United States affecting approximately 100,000 individuals primarily of African ancestry. Pain is the most common complication of SCD. Currently, the mainstay therapy for pain in SCD is opioids. The CDC recommends using non-opioid, non-pharmacologic therapies for pain. There is a growing body of literature to support the use of various integrative therapies for pain.

Acupuncture therapy is a non-pharmacological Chinese medicine approach which has been used in many non-SCD conditions associated with pain. Proposed study will test acceptability and feasibility of use of acupuncture in SCD patients hospitalized for pain. It is hypothesized that the use of acupuncture as an adjuvant therapy will be acceptable to SCD patients admitted for pain control. Its impact on opioid use and circulating cytokines and neuropeptides will also be determined.

DETAILED DESCRIPTION:
This study will evaluate the acceptability and tolerability of acupuncture in patients with SCD admitted for management of acute pain. SCD patients admitted for pain control will be approached for the study. The participants agreeing to receive acupuncture will receive acupuncture once daily for upto 5 days or the day of discharge.

For the primary endpoint of the study, the investigators will determine the proportions of eligible patients/families that are willing to accept acupuncture with their standard of care management of pain. The investigators anticipate ≥60% of patients will agree to accept acupuncture as part of their inpatient pain management.

The investigators also aim to explore whether the use of acupuncture affects opioid use during hospitalization. This secondary endpoint will evaluate opioid use in morphine milligram equivalent (MME) while hospitalized and other outcomes (side effects, pain control and function) which will be compared between the following two groups of patients

1. Treatment group: Participants with SCD hospitalized for acute pain who agree to receive acupuncture (standard of care treatment plus acupuncture)
2. Control group: Participants with SCD hospitalized for acute pain who decline to receive acupuncture (standard of care treatment alone) but agree to serve as controls to allow the study team to collect data on pain-related outcomes (secondary end-points above).

This study will also explore if acupuncture modifies the concentration of circulating cytokines and neuropeptides in the study participants. The study team will draw blood at baseline before acupuncture treatment and on the day of discharge or when the decision to discharge to home will be made by the inpatient team. Concentrations of circulating cytokines and neuropeptides will be compared between the groups. .

ELIGIBILITY:
Inclusion Criteria:

* subjects with SCD (HbSS, HbSC, HbSβ0 thalassemia, HbSOArab)
* Admitted for management of pain at Children's National.
* Ability to provide informed consent/assent

Exclusion Criteria:

* Inability to give informed consent/assent as determined by the investigators
* SCD related complications such as acute chest syndrome requiring supplemental oxygen, fever with bacteremia or concern for serious infection ex. osteomyelitis Local -skin infection or condition not feasible for acupuncture
* Pregnancy or lactation

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Recruitment ratio | Duration of the study upto 5 years
  Number of participants with SCD hospitalized for acute pain who enroll in the study on the acupuncture arm /total number of SCD patients hospitalized for acute pain who enroll in the study will be assessed. This information will determine if acupuncture is a acceptable treatment modality for patients with SCD hospitalized for pain.

SECONDARY OUTCOMES:
Opioid use in morphine milligram equivalents (MME) | Duration of hospitalization up to 5 days
  Opioid use in MME will be calculated in both group of study participants (acupuncture with standard of care arm and standard of care arm) to determine if there are any difference in opioid use between the groups.

OTHER OUTCOMES:
Concentration of circulating cytokines and neuropeptides | Duration of hospitalization up to 5 days
  Circulating cytokines and neuropeptide will be measured in the participants of both groups (acupuncture with standard of care arm and standard of care arm) at baseline and on discharge or day 5 whatever occurs first to determine if there are any differences in concentration of circulating cytokines and neuropeptides between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Darbari, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Reece-Stremtan S, Mahmood L, Margulies S, Martin B, Rohatgi R, Idiokitas R, Cohen IT, Zhang A, Thaniel L, Hardy SJ, Darbari DS. Acupuncture as an Adjunctive Treatment for Pain in Hospitalized Children With Sickle Cell Disease. J Pain Symptom Manage. 2021 Dec;62(6):1239-1244. doi: 10.1016/j.jpainsymman.2021.06.003. Epub 2021 Jun 9. PMID 34118373